CLINICAL TRIAL: NCT01015261
Title: Comparison of Efficacy of Allogenic Bone Marrow Transplantation With Cytoreduction and Chemotherapy in ALL Patients
Brief Title: Allogenic Bone Marrow Transplantation (BMT) Compare With Cytoreduction and Chemotherapy in Acute Lymphoblastic Leukemia (ALL) Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Mahdi Jalili MD / Hematology-Oncology and SCT Research Center, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HORCSCT-0903
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL; BMT; Chemotherapy; Allogenic
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bone Marrow Transplantation; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone Marrow Transplantation (Experimental)
  Interventions: Procedure: Bone Marrow Transplantation
- Chemotherapy (Active Comparator)
  Interventions: Procedure: Chemotherapy

INTERVENTIONS:
Procedure: Bone Marrow Transplantation — Allogenic Bone Marrow Transplantation
  Arms: Bone Marrow Transplantation
Procedure: Chemotherapy — 1. Cyclophosphamide 1200 mg/m2 D15
  2. Daunorubicin 45 mg/m2 D15-D18
  3. Vincristine 1 mg/m2 D15, D22
  4. Dexamethasone 24 mg/d D12-D28
  Arms: Chemotherapy

SUMMARY:
Patients with newly diagnosed Acute lymphoblastic leukemia after providing consent, will be screened for eligibility. Eligible patients will be treated with Vincristine (1 mg/m2 at Day 1 and Day 8), Dexamethasone 24 mg/d day 1-15 and IT at Days 1, 4, 8 and 12. At day 14 patients will be randomized in two group. BMT group who have donor and Chemotherapy group who don't have suitable donor. BMT group treated with allogenic Bone Marrow Transplantation and Chemotherapy treated with Cyclophosphamide at day 15, Daunorubicin at day 15-18, Vincristine at day 15 and 22 and Dexamethasone at day 12-28 followed by standard chemotherapy. In BMT group patients will be received CNS radiotherapy at +100 day after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of Acute lymphoblastic leukemia
* Age between 16 to 50 year
* New case of ALL

Exclusion Criteria:

* Primary CNS involvement
* Primary Testis involvement
* Previously treated

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of allogenic BMT compare with cytoreduction and chemotherapy in ALL patient | 1 year

SECONDARY OUTCOMES:
Overall Survival after BMT compare with chemotherapy. | 1 year
Disease Free Survival after BMT compare with chemotherapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ardeshir Ghavamzadeh, MD, Study Chair — Hematology-Oncology and SCT Research Center
Locations (1):
- Hematology-Oncology & SCT Research Center, Tehran, Tehran Province, Iran